CLINICAL TRIAL: NCT01881256
Title: The BabyGrow Longitudinal Study of Nutrition and Growth in Preterm Infants
Acronym: BabyGrow
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Mairead Kiely, Dr, University College Cork
Other Study IDs: BabyGrow1 Study
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Premature Birth of Newborn; Malnutrition; Intrauterine or Fetal, Small-for-dates
Keywords: Preterm birth; Parenteral and enteral nutrition; Body composition in preterm infants
MeSH Terms: conditions — Premature Birth; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a longitudinal, observational study on nutrition, growth and body composition in preterm infants. Aims to determine the adequacy of actual nutrient intake during the preterm period by investigating associations between macronutrient supply, growth, and body composition at 34-weeks gestation, term equivalent and 2-month corrected gestational age.

DETAILED DESCRIPTION:
Infants between 23 and 24 weeks gestation and with a birth weight of 500 to 1500 g are recruited to a longitudinal, observational study of nutrition, growth and body composition in Cork University Maternity Hospital, Ireland.

ELIGIBILITY:
Inclusion Criteria:

* Babies with a birth weight ≤1.5kg and gestational age ≤34 weeks were considered eligible.

Exclusion Criteria:

* presence of congenital abnormalities or conditions that interfere with growth or body composition (congenital diseases, chromosomal abnormalities, chronic lung disease, cardiac or gastrointestinal diseases).

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants admitted to Cork University Maternity Hospital Neonatal Unit
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Actual nutrient intake vs recommended nutrient requirements in preterm infants | 19 months
  Comparison of intake with requirements during the preterm infant's hospital stay and up to 2 months corrected gestational age.

SECONDARY OUTCOMES:
Longitudinal data on body composition in Irish preterm neonates | 19 months
  Evaluation of appropriateness of current feeding regimens for achievement of optimal growth & body composition outcomes
Longitudinal data on vitamin D intake and circulating 25(OH)D | 19 months
  To examine the relationship between vitamin D intake and serum 25-hydroxyvitamin D concentrations and biomarkers of calcium handling by analysis of sequential serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Mairead E Kiely, PhD, Principal Investigator — University College Cork